CLINICAL TRIAL: NCT07098572
Title: Efficacy of EMG-triggered Four-Channel Functional Electrical Stimulation vs. Cyclic One-Channel Electrical Stimulation on Moderate Arm/Hand Paresis in Subacute Stroke Patients. A Randomized Controlled Single Blinded Multicenter Study
Brief Title: Comparison of Four-Channel Functional Electrical Stimulation vs. One-Channel Electrical Stimulation on Moderate Arm/Hand Paresis in Subacute Stroke Patients
Acronym: MKES2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MED-EL_CRD_2024_02
Record Dates: First submitted 2025-07-24; First posted 2025-08-01 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Moderate Arm Paresis; Ischemic Stroke
Keywords: Arm Paresis; Hand Paresis; Stiwell Profes; Electrostimulation; Ischemic stroke; Rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclic Neuromuscular Electrical Stimulation (cNMES) (Active Comparator): Single channel cyclic neuromuscular stimulation used for the rehabilitation of moderate arm paresis
  Interventions: Device: Cyclic single channel neuromuscular stimulation
- Electromyographic-triggered Multichannel Electrical Stimulation (EMG-MES) (Experimental): EMG-triggered, four channel neuromuscular stimulation used for the rehabilitation of moderate arm paresis
  Interventions: Device: Electromyogram-triggered 4 channel neuromuscular stimulation

INTERVENTIONS:
Device: Cyclic single channel neuromuscular stimulation — Cyclic single channel neuromuscular stimulation is used to trigger repetitive muscular contractions
  Arms: Cyclic Neuromuscular Electrical Stimulation (cNMES)
Device: Electromyogram-triggered 4 channel neuromuscular stimulation — EMG-MES provides biofeedback by using electromyographic signals to trigger muscular contractions
  Other Names: EMG-MES
  Arms: Electromyographic-triggered Multichannel Electrical Stimulation (EMG-MES)

SUMMARY:
This study will compare two treatments that may help participants recover after having suffered from stroke. Persons who experience weakness or paralysis of their arms/hands will be randomly placed in one of two groups. Each receives treatment five times a week for three weeks. One group will be treated with electrostimulation following a cyclic pattern (control treatment), the other group will be treated with electrostimulation triggered by nerve signals (i.e. stimulation starts when they deliberately try to move their arm (investigational treatment). Before and after the three weeks and additionally 12 weeks later, the ability to move the arm and hand will be documented with standardized tests.

ELIGIBILITY:
Inclusion Criteria:

* First-time ischemic stroke with moderate arm paresis (Motricity Index - UE Sum-Score ≥ 40 ≤ 77 points) (Collin & Wade, 1990)
* Early to late subacute phase (7 days - 6 months) (Bernhardt et al., 2017)
* Existing ADL ability before the event (ICF d5 self-care, d6 domestic life, extent of problem ≤1 points) (WHO, 2001)
* Age ≥18 - 99 years
* Signed and dated ICF before the start of any study-specific procedure.

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Implanted defibrillators, brain stimulators, pacemakers, medication pumps
* Therapy-resistant epilepsy
* Fever or infectious diseases
* Inflammatory or tumorous skin diseases in the stimulation area,
* Thromboses or vein inflammations
* Severe contractures of the affected extremity
* Wounds in the stimulation area
* Pregnancy
* Known allergic reactions to components of the investigational medical device
* Unstable psychological status
* Participation in other pharmacological clinical investigations within four weeks prior to enrolment
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale (SIS) subscale Recovery | pre-intervention to 3 weeks
  Scores between 0 and 100, higher meaning a better outcome

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS), subscale strength | pre-intervention to 3 weeks
  Scores between 0 and 100, higher meaning a better outcome
Stroke impact scale (SIS) subscale Activities of Daily Living (ADL) / Instrumental Activities of Daily Living (IADL) | pre-intervention to 3 weeks
  Scores between 0 and 100, higher meaning a better outcome
Stroke impact scale (SIS) subscale mobility | pre-intervention to 3 weeks
  Scores between 0 and 100, higher meaning a better outcome
Stroke impact scale (SIS) subscale hand function | pre-intervention to 3 weeks
  Scores between 0 and 100, higher meaning a better outcome
Fugl-Meyer Assessment - upper extremity (FMA-UE) | pre-intervention to 3 weeks
  Scores between 0 and 100, higher meaning a better outcome
Action Research Arm Test (ARAT) | pre-intervention to 3 weeks
  Scores between 0 and 57, higher meaning a better outcome
Safety assessment | through study completion, an average of 15 weeks
  Assessment of device related adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - KABEG Gailtal-Klinik LKH Hermagor, Hermagor, Carinthia
  - Ö. Landeskrankenhaus Hochzirl - Natters, Standort Hochzirl, Zirl, Tyrol
  - Kepler Universitätsklinikum Linz, Linz, Upper Austria

IPD SHARING:
Plan to Share IPD: Undecided